CLINICAL TRIAL: NCT06959888
Title: A Phase 1 Study in Healthy Volunteers to Evaluate the Relative Bioavailability of ALG-055009 Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aligos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ALG-055009-304
Record Dates: First submitted 2025-03-24; First posted 2025-05-07 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteer Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A (Experimental): Single dose PO administration of 0.7 mg ALG-055009 (Formulation 1; Day 1), then a washout period of at least 7 days, followed by single dose PO administration of 0.7 mg ALG-055009 (Formulation 2; Day 8)
  Interventions: Drug: ALG-055009
- Sequence B (Experimental): Single dose PO administration of 0.7 mg ALG-055009 (Formulation 2; Day 1), then a washout period of at least 7 days, followed by single dose PO administration of 0.7 mg ALG-055009 (Formulation 1; Day 8)
  Interventions: Drug: ALG-055009

INTERVENTIONS:
Drug: ALG-055009 — Single PO dose of 0.7 mg ALG-055009 softgel capsule (formulation 1)
  Single PO dose of 0.7 mg ALG-055009 softgel capsule (formulation 2)

SUMMARY:
This is a phase 1 single dose, open-label, randomized, two-period, two-sequence, crossover study of ALG-055009 conducted in 1 cohort of healthy volunteers. The primary purpose of this study is to compare the single-dose pharmacokinetics of the 0.7 mg dose level of 2 types of soft gelatin capsule formulations of ALG-055009, Formulation 1 and Formulation 2, in approximately 8 healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must sign an informed consent form (ICF) indicating that he or she understands that risks of purpose of and procedures required for, the study and is willing to participate in the study.
2. In the investigator's opinion, the subject is able to understand and comply with protocol requirements, instructions, and protocol stated restrictions and is likely to complete the study as planned.
3. Male or female between 18 and 65 years of age, extremes included.
4. Subjects must have a bod mass index (BMI) of 18.0 to 32.0 kg/m2, extremes included.
5. Female subjects must be either:

   1. Post menopausal: A postmenopausal state is defined as no menses for at least 12 months without an alternative medical explanation . A high follicle-stimulating hormone (FSH) level in the postmenopausal range of >40 IU may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy (HRT).

      OR
   2. Permanently Sterile : Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.

      OR
   3. Woman of Childbearing Potential: They are only eligible if they and any non-sterile male sexual partners agree to use highly effective contraceptive therapy from the screening visit until at least 60 days after the last dose of study drug
6. Female subjects must have a negative pregnancy test at screening and Day-1.
7. Female subjects must not be pregnant, or breastfeeding, or planning to become pregnant or donate eggs from screening onward until 60 days after the last dose of study drug (or longer if dictated by local regulation).
8. Male subjects must agree to wear a condom during sexual intercourse and their female sexual partners should agree to use effective means of contraception. These contraceptive measures must be implemented, at a minimum, from the start of dosing until at least 90 days after the last dose.
9. Male subjects must have no plans to father a child or donate sperm while enrolled in this study or within 90 days after the last dose of study drug.
10. Subjects must have a 12-lead ECG that meets the following inclusion criteria

    1. Heart rate between 40 and 100 beats per minute (bpm), extremes included;
    2. QT interval corrected for heart rate (QTc) according to Fridericia's formula (QTcF) ≤450 ms (males) or ≤470 ms (females);
    3. QRS interval ≤120 ms;
    4. PR interval ≤110 to ≤220 ms;
    5. In addition to fulfilling the above ECG criteria, ECG morphology must have no clinically significant abnormalities observed in the opinion of the Investigator.
11. Subjects must be deemed to be in good overall health by the investigator on the basis of a medical evaluation that reveals the absence of any clinically significant abnormality and includes a physical examination, medical history, vital signs, and the results of blood chemistry, blood coagulation and hematology tests, and a urinalysis performed at screening.
12. Subjects must be willing and able to adhere to the prior and concomitant medications requirements

Exclusion Criteria:

Any potential subject who meets any of the following criteria will be excluded from participating in the study.

1. Subjects with any current or previous illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject or that could prevent, limit, or confound the protocol specified assessments or study results' interpretation. This may include, but is not limited to renal, cardiac, vascular, pulmonary, gastrointestinal, hepatologic, endocrine, neurologic, dermatologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances.
2. Subjects with medical history or current evidence of a pituitary disorder or thyroid disorder.
3. Subjects with thyroid-stimulating hormone (TSH), free thyroxine (T4) or total triiodothyronine
4. Subjects with known sensitivity to thyroid medications
5. The laboratory values at screening are exclusionary:

   1. ALT or AST > ULN
   2. Total bilirubin > 1.2xULN, unless Gilbert's syndrome is suspected
6. Subjects with a past history of cardiac arrhythmias, risk factors for Torsade de Pointes syndrome (e.g., hypokalemia, family history of long QT syndrome ) or history or clinical evidence at screening of significant or unstable cardiac disease, such as: angina, congestive heart failure, myocardial infarction, diastolic dysfunction, significant arrhythmia.
7. History of unexplained syncope.
8. Subjects with current:

   1. Hepatitis A virus infection (confirmed by hepatitis A antibody immunoglobulin M [IgM]).
   2. Hepatitis B infection defined as presence of HBsAg or HBV core antibody.
   3. Hepatitis C virus (HCV) infection (confirmed by HCV antibody and/or HCV RNA). Subjects who have been treated and achieved sustained virologic response ≥6 months prior to screening with HCV RNA <LLOQ, target not detected, remain eligible.
   4. Human immunodeficiency virus type 1 (HIV-1) or HIV-2 infection (confirmed by antibodies) at screening.
   5. Acute infection at the time of enrollment. If an acute infection is considered resolved prior to enrollment, the subject remains eligible.
9. Subjects who had major surgery (e.g., requiring general anesthesia) within 12 weeks before randomization, or will not have fully recovered from surgery, or have surgery planned during the time the subjects is expected to participate in the study, or within 4 weeks after the last dose of study drug
10. Subjects with a recent (within 1 year of randomization/enrollment) history of use of amphetamines, barbiturates, narcotic or other drugs of abuse/recreational drug use. Use of these drugs under physician supervision (e.g., prescription narcotics for known pain disorder) are not exclusionary. Cannabis use within 4 weeks of screening and during the study is exclusionary.
11. Excessive use of alcohol defined as regular consumption of ≥14 standard drinks/week for women and ≥21 standard drinks/week for men (Chalasani et al. 2018). For current definition of a standard drink, please refer to the National Institute on Alcohol Abuse and Alcoholism website (https://www.niaaa.nih.gov/what-standard-drink).
12. Unwilling to abstain from alcohol use for 48 hours prior to Day -1 through end of study follow up.
13. Positive results for urine drug screen or alcohol test at screening or Day -1.
14. Any laboratory result considered clinically significant by the Investigator at screening. Values of ALT and AST >ULN, and total bilirubin >1.2×ULN (see Exclusion Criteria 6), and values of TSH, free T4, and total T3 >1.1×ULN and <0.9×LLN (see Exclusion Criteria 4) are exclusionary regardless of any clinical significance assessment by the Investigator.
15. Clinically significant abnormal vital signs (evaluated in the semi-recumbent [i.e., elevation of the head-to-bed at 30-45 degrees] or supine position after 5 minutes of rest), confirmed with retesting after at least 5 minutes of additional rest. Vital sign reference ranges to assess eligibility are as follows:

    1. Systolic blood pressure: ≥90 to ≤140 mmHg
    2. Diastolic blood pressure: ≥40 to ≤90 mmHg
    3. Pulse rate: ≥40 to ≤100 beats per minute
16. Physical examination findings that are considered clinically significant and likely to adversely impact study conduct and/or interpretation are exclusionary.
17. Renal dysfunction [e.g., estimated creatinine clearance <90 mL/min/1.73 m2 at screening, calculated by the 2021 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula (without correction for African ancestry)].
18. History of clinically significant drug allergy such as, but not limited to, sulfonamides or drug allergy witnessed in previous studies with experimental drugs.
19. Has taken or requires treatment with: any therapies as noted in Prior and Concomitant Medications (Section 6.10) and Special Precautions (Section 6.11) within 1 week or 5 half-lives (whichever is longer) before the planned first dose of study drug or during dosing; any Prohibited Medications (Appendix B) within 28 days or 5 half-lives (whichever is longer) before the planned first dose of study drug or during dosing.
20. Consumption of grapefruit, grapefruit juice, and Seville oranges within 14 days prior to study drug administration.
21. Consumption of apple or orange juice, citrus fruits, vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard), and charbroiled meats within 7 days prior to study drug administration.
22. Consumption of any food or drink/beverage containing quinine (e.g., tonic, bitter lemon, bitter alcoholic beverages containing quinine) within 24 hours prior to study drug administration.
23. Received an unapproved investigational agent within 4 weeks (or 5 half-lives, whichever is longer) prior to enrollment.
24. Currently participating in another clinical or medical interventional research study.
25. Employee of the Sponsor, the Investigator or study site, with direct involvement in the proposed study or other studies under the direction of that Investigator or study site, as well as family members of the employees or the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
AUC0-24 of ALG-055009 in Plasma | 12 days
  AUC0-24, of ALG-055009 in plasma following single dose administration of 0.7 mg ALG-055009 Formulation 1 and Formulation 2
AUClast of ALG-055009 in Plasma | 12 days
  AUClast of ALG-055009 in plasma following single dose administration of 0.7 mg ALG-055009 Formulation 1 and Formulation 2
AUCinf of ALG-055009 in Plasma | 12 days
  AUCinf of ALG-055009 in plasma following single dose administration of 0.7 mg ALG-055009 Formulation 1 and Formulation 2
Tmax of ALG-055009 in Plasma | 12 days
  Tmax of ALG-055009 in plasma following single dose administration of 0.7 mg ALG-055009 Formulation 1 and Formulation 2
Cmax of ALG-055009 in Plasma | 12 days
  Cmax of ALG-055009 in plasma following single dose administration of 0.7 mg ALG-055009 Formulation 1 and Formulation 2
C24 of ALG-055009 in Plasma | 12 days
  C24 of ALG-055009 in plasma following single dose administration of 0.7 mg ALG-055009 Formulation 1 and Formulation 2
C0 (predose) of ALG-055009 in Plasma | 12 days
  C0 (predose) of ALG-055009 in plasma following single dose administration of 0.7 mg ALG-055009 Formulation 1 and Formulation 2
t½ of ALG-055009 in Plasma | 12 days
  t½ of ALG-055009 in plasma following single dose administration of 0.7 mg ALG-055009 Formulation 1 and Formulation 2

SECONDARY OUTCOMES:
Safety Data | 22 days
  The number and severity of treatment emergent adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Austin CRU, Austin, Texas, United States